CLINICAL TRIAL: NCT05489653
Title: Effects of Mixed Music Intervention on Improving Sleep Disturbance in Patients With Parkinson's Disease: a Feasibility Randomized Controlled Trial
Brief Title: Mixed Music Intervention on Sleep Disturbance in Patients With Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting cases due to the epidemic
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202204014
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Music Intervention; Sleep Disturbance; Parkinson's Disease
MeSH Terms: conditions — Parasomnias; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mixed music group (Experimental): If assigned to the mixed music group, in order to synchronize active daytime music and passive music at bedtime, active daytime music will require patients to perform physical music activities once a week and watch a recorded music intervention video three times a week during the study period (The content is the same as the physical music activities) and follow the activities, and the intervention content before going to bed is the same as the intervention content of the pure passive music group.
  Interventions: Behavioral: mixed music
- pure passive music group (Active Comparator): If assigned to the pure passive music group, they are required to listen to soft and low-pitched music at about 60 beats per minute 30 minutes before bed every day for four weeks.
  Interventions: Behavioral: mixed music
- conventional treatment (No Intervention): Conventional treatment group maintained their original lifestyle and were post-tested with the assistance of a single-blind study evaluator.

INTERVENTIONS:
Behavioral: mixed music — Learn about the effects of listening to music and doing activities with it on sleep.
  Arms: mixed music group; pure passive music group

SUMMARY:
Parkinson's disease is a disease that is prevalent in the elderly, and the risk increases with age. Sleep disturbance is a common complaint of patients with Parkinson's disease, with a prevalence of 60% to 96%. Long-term sleep disturbance in Parkinson's disease patients significantly reduces cognitive function and quality of life. Nursing staff are the first line of care and should seek appropriate strategies to address sleep disturbances in patients with Parkinson's disease.

This study is a feasibility and pilot study, which will be a single-blind, parallel randomized controlled trial. It is expected to include 30 patients with Parkinson's disease with poor sleep quality, and they will be equally allocated to the mixed music group (10 people), passive music group (10 people), and usual care group (10 people) in a 1:1:1 ratio. If assigned to the passive music group, they are required to listen to soft and low-pitched music at about 60 beats per minute for 30 minutes before sleep every day for four weeks. If assigned to the mixed music group, in order to synchronize active daytime music and passive music at bedtime, active daytime music will require patients to perform physical music activities once a week and watch a recorded music intervention video three times a week during the study period (The content is the same as the physical music activities) and follow the activities, and the intervention content before going to bed is the same as the intervention content of the pure passive music group. Subjects assigned to the usual care group maintained their original lifestyle and were assisted by study evaluators to complete pre-and post-test data. The researchers will establish a line group, and the three groups of patients or primary caregivers will be contacted by line every two days to care for the patient's condition. The variables measured included anxiety, depression, quality of life, and sleep quality, as assessed by the Hospital Anxiety and Depression Scale, Parkinson 's Disease. Questionnaire - 39, and the Pittsburgh Sleep Quality Scale . This study will use one-way ANOVA and linear mixed model for statistical analysis to test the hypothesis of this study.

If the effectiveness of this intervention can be confirmed, it will be implemented in Parkinson's disease patients in the future to reduce sleep disturbances and improve patients' quality of life.

DETAILED DESCRIPTION:
Parkinson's disease is a disease that is prevalent in the elderly, and the risk increases with age. Sleep disturbance is a common complaint of patients with Parkinson's disease, with a prevalence of 60% to 96%. Long-term sleep disturbance in Parkinson's disease patients significantly reduce cognitive function and quality of life. Nursing staff are the first line of care and should seek appropriate strategies to address sleep disturbances in patients with Parkinson's disease. In the past, it has been pointed out that passive music therapy can improve sleep disorders, but there is no active music intervention to improve sleep disorders in Parkinson's disease patients, and there is no combination of active and passive music intervention to improve the sleep disorders of this group. Therefore, this study will investigate the effect of active and passive music intervention in improving sleep disturbance in Parkinson's disease patients in a randomized controlled trial.

The purpose of this study was to investigate the effect of active and passive music intervention in improving sleep disturbance in Parkinson's disease patients. This study assumes that active and passive music interventions are feasible intervention measures. Compared with passive music intervention and conventional treatment, active combined passive music intervention is expected to improve the sleep quality and quality of life of patients with Parkinson's disease.

This study is a feasibility and pilot study, which will be a single-blind, parallel randomized controlled trial. It is expected to include 30 Pittsburgh patients with Parkinson's disease with a sleep quality expression of more than 5 points , and they will be equally allocated to the mixed music group (10 people), the pure passive music group (10 people) and conventional treatment in a 1:1:1 ratio. Group (10 people). If assigned to the pure passive music group, they are required to listen to soft and low-pitched music at about 60 beats per minute 30 minutes before bed every day for four weeks. If assigned to the mixed music group, in order to synchronize active daytime music and passive music at bedtime, active daytime music will require patients to perform physical music activities once a week and watch a recorded music intervention video three times a week during the study period (The content is the same as the physical music activities) and follow the activities, and the intervention content before going to bed is the same as the intervention content of the pure passive music group. Subjects assigned to the usual care group maintained their original lifestyle and were assisted by study evaluators to complete pre-and post-test data. The researchers will establish a line group, and the three groups of patients or primary caregivers will be contacted by line every two days to care for the patient's condition. The variables measured included anxiety, depression, quality of life, and sleep quality, as assessed by the Hospital Anxiety and Depression Scale, Parkinson 's Disease. Questionnaire - 39, and the Pittsburgh Sleep Quality Scale . This study will use one-way ANOVA and linear mixed model for statistical analysis to test the hypothesis of this study.

If the effectiveness of this intervention can be confirmed, it will be implemented in Parkinson's disease patients in the future to reduce sleep disturbances and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The test subjects must be adults or elderly aged 30 to 80 years old, with clear consciousness (Glasgow Coma Scale score 15), no obvious hearing impairment, diagnosed with Parkinson's disease in the first to third stages, Pittsburgh sleep quality expression is more than 5 points, has the ability to move independently with assistance,can communicate in Chinese or Taiwanese, and usually be accompanied by the main caregiver or family members.

Exclusion Criteria:

* Exclusions included skeletal injuries or medical orders that restricted or prohibited activities prior to the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | four-week intervention
  Sleep quality will be assessed by the Chinese version of the Pittsburgh Sleep Quality Scale, which is divided into subjective sleep quality, sleep quality and sleep quality. Lag period, total sleep hours, habitual sleep efficiency, sleep disturbance, sleep medication use, and daytime functional status.
  The total Pittsburgh sleep quality index is the total score of the seven major parts, so the total score is up to 21 points. If the total score is more than 5 points, it means sleep The quality is not good; on the contrary, the total score is ≤ 5 points, which means the sleep quality is good. Chinese version of Pittsburgh Sleep Quality Scale Internal Consistency (Cronbach's alpha) ranged from 0.82 to 0.83, with a sensitivity and specificity of 98% and 55%. Therefore, the scale is an accurate and reliable assessment tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No